CLINICAL TRIAL: NCT04609475
Title: Osseodensification Versus Motor-Driven Expanders' Techniques for Increasing Bone Density With Simultaneous Implant Placement (Randomized Controlled Clinical Trial)
Brief Title: Osseodensification Versus Motor-Driven Expanders' Techniques for Increasing Bone Density With Simultaneous Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Osseodensification technique
Record Dates: First submitted 2020-10-24; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Alveolar Bone Loss
Keywords: Endosseous implants; Osseodensification
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osseodensification technique (Experimental)
  Interventions: Procedure: Osseodensification technique
- Motor driven expanders' technique (Active Comparator)
  Interventions: Procedure: Motor driven expanders' technique

INTERVENTIONS:
Procedure: Osseodensification technique — Implant bed preparation will be performed according to the manufacturer's guidelines, densifying burs (Densah® Burs) will be used sequentially in densifying mode (counterclockwise drill speed 800-1500 rpm with copious irrigation) to achieve the planned osteotomy diameter and desired ridge expansion. The implant will be then placed in the prepared osteotomy
  Arms: Osseodensification technique
Procedure: Motor driven expanders' technique — The technique consisted of preparing the implant bed by progressively increasing the size of the osteotomes until the desired expansion will be achieved. At the planned implant site, a pilot drill 1000 rpm with irrigation until the desired length, then expansion with the series of ridge spreaders and finally using the final drill. The implant will be then placed in the prepared osteotomy.
  Arms: Motor driven expanders' technique

SUMMARY:
The aim of this study was to compare and measure the amount of bone density and ridge width gained with motor driven expanders and densifying burs with simultaneous dental implant placement.

DETAILED DESCRIPTION:
Seven patients were treated by the osseodensification technique and another seven were treated by the motor-driven expanders' technique with simultaneous implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring implant placement in the anterior maxilla until the premolar region.
* Patients are medically fit.
* The width of the deficient maxillary alveolar ridge not less than 3mm.
* Patients willing and fully capable to comply with the study protocol.

Exclusion Criteria:

* Atrophic ridge (2 mm or less) with no interposition of cancellous bone between the buccal and palatal plates.
* Uncontrolled metabolic disease (e.g. uncontrolled diabetes).
* Heavy smokers (>15 cigarettes/day).
* Acute oral infections.
* Untreated periodontal disease.
* Poor oral hygiene.
* Pregnant or breastfeeding patient.
* A history of radiotherapy to the head and neck region or treatment with bisphosphonates.
* Female patients using oral contraceptive pills.
* Presence of oral parafunctional habits.
* Surgical site needs to be grafted.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | up to 1 month
  Pain was assessed using a 10-point Visual Analogue Scale (VAS). The lower values indicates lower pain levels and higher values indicates higher pain levels
Implant stability | up to 6 months
  Stability was assessed using resonance frequency analysis measured with the Osstell device instrument. The Osstell unit records a numeric value of 1-100 which is referred to as the implant stability quotient (ISQ). The measurements were performed and 3 mean of three readings were recorded.
Bone density | up to 6 months
  This will be assessed using cone beam computed tomography (CBCT)

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa A Abdou, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Magued H Fahmy, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Ahmed O Sweedan, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Alghamdi H, Anand PS, Anil S. Undersized implant site preparation to enhance primary implant stability in poor bone density: a prospective clinical study. J Oral Maxillofac Surg. 2011 Dec;69(12):e506-12. doi: 10.1016/j.joms.2011.08.007. PMID 22117707
- [Background] Boustany CM, Reed H, Cunningham G, Richards M, Kanawati A. Effect of a modified stepped osteotomy on the primary stability of dental implants in low-density bone: a cadaver study. Int J Oral Maxillofac Implants. 2015 Jan-Feb;30(1):48-55. doi: 10.11607/jomi.3720. PMID 25615915
- [Background] Bornstein MM, Cionca N, Mombelli A. Systemic conditions and treatments as risks for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:12-27. PMID 19885432
- [Background] Hatano N, Shimizu Y, Ooya K. A clinical long-term radiographic evaluation of graft height changes after maxillary sinus floor augmentation with a 2:1 autogenous bone/xenograft mixture and simultaneous placement of dental implants. Clin Oral Implants Res. 2004 Jun;15(3):339-45. doi: 10.1111/j.1600-0501.2004.00996.x. PMID 15142097
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329
- [Background] Hwang D, Wang HL. Medical contraindications to implant therapy: Part II: Relative contraindications. Implant Dent. 2007 Mar;16(1):13-23. doi: 10.1097/ID.0b013e31803276c8. PMID 17356368
- [Background] Jimbo R, Tovar N, Marin C, Teixeira HS, Anchieta RB, Silveira LM, Janal MN, Shibli JA, Coelho PG. The impact of a modified cutting flute implant design on osseointegration. Int J Oral Maxillofac Surg. 2014 Jul;43(7):883-8. doi: 10.1016/j.ijom.2014.01.016. Epub 2014 Feb 28. PMID 24583140
- [Background] Johnson C. Measuring Pain. Visual Analog Scale Versus Numeric Pain Scale: What is the Difference? J Chiropr Med. 2005 Winter;4(1):43-4. doi: 10.1016/S0899-3467(07)60112-8. PMID 19674646